CLINICAL TRIAL: NCT00098852
Title: A Pilot Study of Rosiglitazone in Patients With Incurable Differentiated Thyroid Cancer
Brief Title: Rosiglitazone in Treating Patients With Locoregionally Extensive or Metastatic Thyroid Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Electron Kebebew, UCSF Helen Diller Family Comprehensive Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000398114; UCSF-03201; UCSF-H28355-22994-01; GSK-UCSF-H28355-22994-01
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2009-01

CONDITIONS: Head and Neck Cancer
Keywords: recurrent thyroid cancer; stage II follicular thyroid cancer; stage IV follicular thyroid cancer; stage II papillary thyroid cancer; stage IV papillary thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Neoplasms; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary | interventions — Rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone maleate

SUMMARY:
RATIONALE: Drugs such as rosiglitazone may make tumor cells more sensitive to radioactive iodine.

PURPOSE: This phase II trial is studying how well rosiglitazone works in treating patients with locoregionally extensive or metastatic thyroid cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine complete response in patients with locoregionally extensive or metastatic differentiated thyroid cancer treated with rosiglitazone.

Secondary

* Compare the long-term response of patients treated with this drug with historical controls.
* Determine the toxicity profile of this drug in these patients.
* Determine the presence/persistence of tumor in patients treated with this drug.
* Determine the quality of life of patients treated with this drug.
* Determine overall survival of patients treated with this drug.

OUTLINE: This is a pilot study.

Patients receive oral rosiglitazone once daily on weeks 1-8. Patients also receive oral liothyronine sodium twice daily on weeks 1-6 in preparation for radioactive iodine scan. Treatment continues in the absence of disease progression or unacceptable toxicity. At week 8, all patients undergo whole body radioactive iodine scan followed by a treatment dose of radioiodine to assess radioiodine uptake by tumor.

Quality of life is assessed at baseline and at the end of study treatment.

Patients are followed at 2 weeks, 1, 4, and 10 months, and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 20-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of differentiated thyroid cancer

  * Locoregionally extensive and/or metastatic disease
  * Inoperable disease
* Failed prior conventional therapy that included total/near-total thyroidectomy AND radioactive iodine I 131 ablation therapy
* Elevated thyroglobulin (Tg) levels (> 3 ng/mL on thyroid hormone OR > 10 ng/mL off thyroid hormone)

  * Tg-antibody positive patients are eligible despite the Tg level
* Radioactive iodine (RAI) scan showing no or therapeutically insignificant (< 1%) RAI uptake after thyroid hormone withdrawal

  * Scan performed within the past 18 months

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 50,000/mm^3

Hepatic

* ALT ≤ 2 times upper limit of normal

Renal

* Creatinine ≤ 1.5 mg/dL

Cardiovascular

* No New York Heart Association class III or IV cardiac disease

Other

* Not pregnant
* No nursing within the past 3 months
* Negative pregnancy test
* Fertile patients must use effective contraception
* No allergy to thiazolidinediones
* No other malignancy except basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 3 months since prior chemotherapy

Endocrine therapy

* See Disease Characteristics
* No concurrent levothyroxine

Radiotherapy

* See Disease Characteristics
* No prior cumulative dose of radioiodine ≥ 800 mCi
* Prior adjuvant or therapeutic external beam radiotherapy allowed

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-10; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Radioiodine uptake and thyroglobulin level at 6 months and 1 year

SECONDARY OUTCOMES:
Side effects of drug at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Electron Kebebew, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States

REFERENCES:
- [Result] Kebebew E, Reiff E, Greenspan FS, et al.: Rosiglitazone treatment induces radioiodine uptake in some patients with radioiodine-negative thyroglobulin-positive differentiated thyroid cancer. [Abstract] The Endocrine Society's 87th Annual Meeting, 4-7 June 2005, San Diego, CA. A-P3-573, 2005. Also available online. Last accessed February 21, 2006.